CLINICAL TRIAL: NCT04765670
Title: Acute Effects of Instrument-assisted Soft Tissue Mobilization and Kinesiotape Application on Pain and Joint Position Sense in Individuals With Chronic Neck Pain.
Brief Title: Instrument-assisted Soft Tissue Mobilization and Kinesiotape Application in Individuals With Chronic Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KaratayUH2
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-02

CONDITIONS: Cervical Pain
Keywords: Chronic cervical pain; Instrument Assisted Soft Tissue Mobilization; Kinesiotape; Joint position sense
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrument Assisted Soft Tissue Mobilization (Experimental): The instruments will be applied to the soft tissue at 30º-60º angles, with multi-directional "stroking" movements. Instrument Assisted Soft Tissue Mobilization will be applied to the trapezius and sternocleidomastoideus muscles of the participants for 90 seconds.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization
- Kinesiotape Application (Experimental): The application will be made from the insertion of the upper trapezoidal muscle to its origo . During taping, the patient will be allowed to sit in an upright position in a chair with a back, with the scapula fixed, without supporting the arms. Before taping, the patient will be positioned with the shoulder in adduction and the head in lateral flexion towards the contralateral side. The patient will be asked to perform shoulder abduction against resistance, and the insertion area of the upper trapezius fibers will be palpated. The initial 2-3 cm part of the band will be glued to the lateral of the acromion without stretching, after full (100%) stretching is applied to the 2-3 cm part of the band from the insertion area of the upper trapezoid fibers, the patient's head is rotated to the affected side and the arm part of the band is stretched along the muscle fibers. it will be glued up to the hairline without doing it.
  Interventions: Other: Kinesiotape Application

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization — Bilateral Instrument assisted soft tissue mobilization application will be applied in a single session to the trapezius and sternocleideomastoideus muscles.
  Arms: Instrument Assisted Soft Tissue Mobilization
Other: Kinesiotape Application — Bilateral Kinesiotape application will be applied in a single session to the trapezius and sternocleideomastoideus muscles.
  Arms: Kinesiotape Application

SUMMARY:
Chronic neck pain causes errors in joint position sense. There are studies in the literature suggesting that instrument-assisted soft tissue mobilization and Kinesiotape applications improve the joint position sense. There is no study examining these applications acutely on joint position sense and pain in the cervical region. As a result of our study, we will compare the effects of single-session instrument-assisted soft tissue mobilization and Kinesiotape application on pain and joint position sense.

DETAILED DESCRIPTION:
The study will be carried out on volunteers after the approval of the ethics committee. Before the research, individuals and / or their relatives will be informed about the purpose and content of the study. Volunteer individuals between the ages of 18-45 with chronic neck pain will be included in the study after obtaining their informed consent.

Participants will be randomly divided into two groups: Instrument assisted soft tissue mobilization and Kinesiotape Applications.

In the instrument-assisted soft tissue mobilization group, the trapezius and sternocleidomastoideus muscles will be applied in a single session for 90 seconds. Kinesiotape application will be applied to the trapezius and sternocleidomastoideus muscles in one session.

Pain will be evaluated with Visual Analog Scale and joint position sense will be evaluated with Cervical Range of Motion device before and after application.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with chronic neck pain
* Being in the age range of 18-45

Exclusion Criteria:

* Those with acute injury or infection,
* Those with open wounds,
* Osteoporosis,
* Hematoma,
* Those with acute cardiac, liver and kidney problems,
* Those with connective tissue disease, Rheumatoid arthritis, osteoarthritis, Cancer,
* Those with circulation problems,
* Those with peripheral vascular disease,
* Epilepsy
* Identified as a history of surgery in the cervical region

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Cervical Pain at 2 minutes | Baseline and 2 minutes after intervention
  Pain will be evaluated with Visual Analog Scale.
Change from Baseline Joint Position Sense at 2 minutes | Baseline and 2 minutes after intervention
  Joint Position Sense will be evaluated Cervical Range of Motion Device

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Gerçek, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)